CLINICAL TRIAL: NCT03886727
Title: Clinical Retention of Bonded Resin Sealants Placed With Rubber Dam Versus Cotton Roll Isolation
Brief Title: Effectiveness of Rubber Dam Isolation Versus Cotton Roll Isolation on Bonded Fissure Sealant Retention
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zafer Cavit Cehreli, DDS, PhD (Other)
Responsible Party: Sponsor-Investigator, Zafer Cavit Cehreli, DDS, PhD, Clinical Professor, Hacettepe University
Organization: Hacettepe University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: RDI vs cotton roll
Record Dates: First submitted 2019-02-21; First posted 2019-03-22 (Actual); Last update posted 2019-11-05 (Actual); Status verified 2019-11

CONDITIONS: Dental Caries in Children; Dental Caries on Pit and Fissure Surface; Dental Leakage
MeSH Terms: conditions — Dental Leakage

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Rubber Dam (Active Comparator): Isolation of single tooth using rubber dam
  Interventions: Device: Rubber Dam Set
- Cotton Roll (Active Comparator): Isolation of quadrant using cotton rolls
  Interventions: Device: Dental Cotton Roll

INTERVENTIONS:
Device: Rubber Dam Set — Rubber dam set is the generic name of an isolation device that consists of a rubber sheet that isolates the tooth from saliva, a clamp to hold the rubber sheet on the tooth to be isolated, and a metal frame to keep the rubber sheet in a stretched position during dental procedures.
  Arms: Rubber Dam
Device: Dental Cotton Roll — Cotton roll is the generic name of a disposable isolation device made of cotton in a cylindrical form. Cotton rolls are used to isolate the teeth from saliva, by being placed in the cheek and tongue during placement of sealants or filings.
  Arms: Cotton Roll

SUMMARY:
The purpose of this study is to evaluate and compare the clinical retention of bonded fissure sealants placed under rubber dam isolation and cotton roll isolation.

ELIGIBILITY:
Inclusion Criteria:

* Teeth having a clinical indication of sealing with bonded resin pit and fissure sealants
* Patients with four fully-erupted permanent molars, with unstained, caries-free and unsealed pit and fissures

Exclusion Criteria:

* Patients having incipient carious lesions, fewer erupted molars or teeth without pits on buccal/palatal surfaces.
* Patients with systemic diseases.

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2020-02-01 (Estimated); Primary Completion 2021-06-01 (Estimated); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
The US Public Health Service criteria for retention of sealants | 12 months
  Alpha: No Loss of sealant, Bravo: Partial Loss of Sealant, Charlie: Total loss of sealant

SECONDARY OUTCOMES:
The US Public Health Service criteria for secondary caries on sealants | 12 months
  Alpha: Charlie: There is no clinical diagnosis of caries. Charlie: There is clinical diagnosis of caries

CONTACTS AND LOCATIONS:
Locations (1):
- LSU School of Dentistry, Department of Pediatric Dentistry, New Orleans, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No